CLINICAL TRIAL: NCT02424357
Title: Suture Contamination Rate in Adjustable Suture Strabismus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Hilda Capo, Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20150111
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Suture Strabismus Surgery
Keywords: Adjustable strabismus surgery; suture contamination; 5%povidone iodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The surgeon will be unaware of the randomization until the end of the surgery. All microbiology personnel and patients will be unaware of the interventional group
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5% povidone iodine ophthalmic solution (Experimental): patient received 1 drop of 5% povidone-iodine instilled over the adjustable suture noose in addition to routine antibiotic/steroid ointment to operated eye at surgery completion
  Interventions: Drug: 5%povidone iodine ophthalmic solution; Drug: routine post-operative ophthalmic ointment
- no povidone-iodine ophthalmic solution (Active Comparator): patient received a routine antibiotic/steroid ointment to operated eye at surgery completion
  Interventions: Drug: routine post-operative ophthalmic ointment

INTERVENTIONS:
Drug: 5%povidone iodine ophthalmic solution — one drop of 5% povidone iodine instilled into the conjunctival fornix.
  Other Names: 5%Betadine ophthalmic drop
  Arms: 5% povidone iodine ophthalmic solution
Drug: routine post-operative ophthalmic ointment — patient received a routine antibiotic/steroid ointment to operated eye at surgery completion

SUMMARY:
1. To establish the culture positivity rate in adjustable suture strabismus surgery
2. To identify bacterial species and antibiotic susceptibility patterns of microorganisms cultured from suture material
3. To compare suture contamination rates with techniques to reduce the suture contamination rate

DETAILED DESCRIPTION:
Patients will be randomized into 1 of 2 groups: those who received 1 drop of 5% povidone-iodine instilled directly over the sliding noose at surgery completion (group 1) and those who did not receive povidone-iodine at the end of the surgery (group 2).

Institutional standard surgical preparation will be performed in all patients with 5% povidone-iodine solution on the periocular skin and eyelid margins, followed by instillation of 1 drop of 5% povidone-iodine into the conjunctival cul-de-sac.

All operations will be performed using a sliding noose technique with a polyglactin 6-0 suture (Vicryl, Ethicon Inc). If a patient undergoes surgery on more than 1 muscle in the same eye, a 1-cm section of suture proximal to the knot will be collected from the nonadjustable suture as a control. The control suture will be placed in a tube with 2 mL of trypticase soy broth and agitated for 1 minute. At the end of surgery, patients in group 1 will receive a drop of povidone-iodine. A strip of neomycin sulfate, polymyxin B sulfate, and dexamethasone ophthalmic ointment will be then applied into the lower conjunctival fornix to patients in both groups.

ELIGIBILITY:
Inclusion Criteria:

* All strabismus patients age ≥ 18 years scheduled for strabismus surgery with adjustable sutures at the Bascom Palmer Eye Institute will be invited to participate.

Exclusion Criteria:

* Patient who has a history of allergy to povidone-iodine.
* Disorders affecting immune function.
* Patient who is unwilling to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hilda Capo, MD, Principal Investigator — Bascom Palmer Eye Institute
Locations (1):
- Bascom Palmer Eye Institute, University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eustis HS, Rhodes A. Suture contamination in strabismus surgery. J Pediatr Ophthalmol Strabismus. 2012 Jul-Aug;49(4):206-9. doi: 10.3928/01913913-20110920-01. PMID 22909077
- [Background] Olitsky SE, Vilardo M, Awner S, Reynolds JD. Needle sterility during strabismus surgery. J AAPOS. 1998 Jun;2(3):151-2. doi: 10.1016/s1091-8531(98)90006-4. PMID 10532751
- [Background] Carothers TS, Coats DK, McCreery KM, Rossman SN, Wilson P, Wu TG, Paysse EA. Quantification of incidental needle and suture contamination during strabismus surgery. Binocul Vis Strabismus Q. 2003;18(2):75-9. PMID 12765540
- [Background] Apt L, Isenberg SJ, Yoshimori R, Chang A, Lam GC, Wachler B, Neumann D. The effect of povidone-iodine solution applied at the conclusion of ophthalmic surgery. Am J Ophthalmol. 1995 Jun;119(6):701-5. doi: 10.1016/s0002-9394(14)72773-4. PMID 7540363
- [Derived] Rossetto JD, Suwannaraj S, Cavuoto KM, Spierer O, Miller D, McKeown CA, Capo H. Evaluation of Postoperative Povidone-Iodine in Adjustable Suture Strabismus Surgery to Reduce Suture Colonization: A Randomized Clinical Trial. JAMA Ophthalmol. 2016 Oct 1;134(10):1151-1155. doi: 10.1001/jamaophthalmol.2016.2926. PMID 27561000

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5% Povidone Iodine Ophthalmic Solution | no Povidone-iodine Ophthalmic Solution
Started | 35 | 30
Completed | 35 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5% Povidone Iodine Ophthalmic Solution | no Povidone-iodine Ophthalmic Solution | Total
Number analyzed (Participants) | 35 | 30 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (16.8) | 46.6 (18.1) | 47.6 (17.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 17 | 10 | 27

OUTCOME MEASURES:

1. Primary Outcome: Suture Colonization Rate in Adjustable Suture Strabismus Surgery
Description: 1 cm section of the suture proximal to the knot will be harvested and placed in a tube with 2 ml of trypticase soy broth (TSB).The TSB tubes will be monitored for growth of bacteria at 48 hours
Time Frame: 48 hours
Measure: Number; unit: percentage sutures positive for bacteria
Units Other Than Participants: sutures
Arm/Group | 5% Povidone Iodine Ophthalmic Solution | no Povidone-iodine Ophthalmic Solution
Number analyzed (Participants) | 35 | 30
Number analyzed (sutures) | 35 | 30
percentage sutures positive for bacteria | 57 | 47

2. Secondary Outcome: Reduction of Contamination Rate Using Post-operative 5% Povidone Iodine
Description: Comparison of suture colonization rates with and without instillation of a drop of povidone-iodine at surgery completion
Time Frame: 48 hours
Measure: Number (95% Confidence Interval); unit: relative risk
Units Other Than Participants: sutures
Groups:
- With or Without 5% Povidone Iodine Ophthalmic Solution: patients with and without 1 drop of 5% povidone-iodine instilled over the adjustable suture noose in addition to routine antibiotic/steroid ointment to operated eye at surgery completion
Arm/Group | With or Without 5% Povidone Iodine Ophthalmic Solution
Number analyzed (Participants) | 65
Number analyzed (sutures) | 65
relative risk | 1.1 [0.6 to 1.7]

3. Secondary Outcome: Identification of Bacterial Species Cultured From Suture Material
Description: The collected sutures will be monitored for bacterial growth for up to 7 days. When bacterial growth is observed, 1 mL of the solution will be inoculated on chocolate, MacConkey, and anaerobic blood agars and incubated for an additional 24 to 48 hours to identify organisms and quantify growth. In vitro susceptibility patterns will be determined.
Time Frame: 7 days plus 24 to 48 hours
Population: All 65 participants were analyzed: 53 sutures had positive cultures (34 of the adjustable sutures and 19 of the control sutures). The relative risk between the two treatment arms indicated no difference in colonization rate, the bacterial species were not analyzed separately. Three of the sutures yielded 2 bacterial species.
Measure: Number; unit: number of positive bacterial isolates
Units Other Than Participants: sutures
Groups:
- With or Without 5% Povidone Iodine Ophthalmic Solution: patients who received 1 drop of 5% povidone-iodine instilled over the adjustable suture noose in addition to routine antibiotic/steroid ointment to operated eye at surgery completion and those that did not receive povidone-iodine
Arm/Group | With or Without 5% Povidone Iodine Ophthalmic Solution
Number analyzed (Participants) | 65
Number analyzed (sutures) | 65
number of positive bacterial isolates
  Staphylococcus epidermidis | 40
  Staphylococcus lugdunensis | 3
  Staphylococcus aureus | 2
  Staphylococcus capitis | 2
  Staphylococcus hominis | 2
  Propionibacterium acnes | 2
  Staphylococcus cohnii | 1
  Staphylococcus warneri | 1
  Staphylococcus xylosus | 1
  Citrobacter koseri | 1
  Lactococcus lactis | 1

ADVERSE EVENTS:
Arm/Group | 5% Povidone Iodine Ophthalmic Solution | no Povidone-iodine Ophthalmic Solution
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/30
Other Adverse Events (participants affected / at risk) | 0/35 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes